CLINICAL TRIAL: NCT02546869
Title: A Single-Arm Study to Evaluate Administration of Lebrikizumab by Participants or Caregivers in the Home Setting
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was withdrawn due to an internal decision.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WB29906
Record Dates: First submitted 2015-09-07; First posted 2015-09-11 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — lebrikizumab

ARMS (1):
- Lebrikizumab (Experimental): Participants will receive lebrikizumab SC using prefilled syringes (PFS), q4w up to Week 12.
  Interventions: Drug: Lebrikizumab; Device: Prefilled Syringes

INTERVENTIONS:
Drug: Lebrikizumab — Lebrikizumab will be administered SC using PFS, q4w up to Week 12.
Device: Prefilled Syringes

SUMMARY:
This multi-center, single-arm study is designed to evaluate clinical experience of participants (or caregivers) administering lebrikizumab at home in participants with asthma. Eligible participants will receive four doses of subcutaneous (SC) lebrikizumab every 4 weeks (q4w) up to Week 12. Primary analysis visit occurs at Week 13. After study treatment, all participants will complete a 12 week safety follow up. All participants will get training for the administartion of lebrikizumab using the device.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 75 years at Week -1
* Asthma diagnosis for greater than or equal to (>=) 12 months prior to Week -1
* Pre-bronchodilator forced expiratory volume in 1 second (FEV1) of >=40% predicted at Week -1 or Week 0 (Day 1; prior to entering treatment phase), based on an established spirometry reference equations
* Competent and willing, as determined by the investigator, to independently administer lebrikizumab at home. The investigator needs to confirm that the participant (or caregiver) will be able to follow the instructions to administer lebrikizumab
* Able and willing to take home the pre-filled syringes of lebrikizumab at the conclusion of Week 0 (Day 1) and store these according to the requirements highlighted within the Instructions for Use (IFU) document.

Exclusion Criteria:

* History of a severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the lebrikizumab injection
* Hospitalization for any reason, including acute exacerbation event, within 4 weeks prior to Week -1 or during the screening period
* Infection that required hopitalization, treatment with intravenous (IV) or intramuscular antibiotics within 4 weeks and oral antibiotics within 2 weeks prior to Week -1 or during screening
* Taken part in a previous clinical trial of lebrikizumab and discontinued from the trial prematurely or discontinued study drug prematurely due to an adverse event

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2016-06-29 (Estimated); Study Completion 2016-06-29 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with adherence to each planned home administration | up to Week 13

SECONDARY OUTCOMES:
Percentage of participants who reported device complaints | up to Week 13
Serum lebrikizumab concentration at Weeks 13 and 24 | Week 13 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche